CLINICAL TRIAL: NCT05697887
Title: Feasibility, Tolerability and Efficacy of the Ketogenic Diet in Children With Drug-resistant Epilepsy in South Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Number 2 Children's Hospital, Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Thuy-Minh-Thu NGUYEN, MD, Number 2 Children's Hospital, Ho Chi Minh City
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH2HCM
Record Dates: First submitted 2022-12-29; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Drug Resistant Epilepsy; Ketogenic Diet; Feasibility; Tolerability; Efficacy; Children
Keywords: drug resistant epilepsy; ketogenic diet
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Children with drug-resistant epilepsy followed at Children's Hospital No.2, Viet Nam treated by KD were included in a prospective study from June 2019 to October 2021. Side-effects, retention rate, number, and duration of seizures were recorded after 1, 3, 6, 9 and 12 months of KD. Patients were considered as responder when a 50% seizure frequency was reached. Tolerance and acceptability of the KD were closely monitored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The feasibility of the ketogenic diet (Experimental): The purpose of this study was to verify the feasibility of the ketogenic diet in children with refractory epilepsies followed at a pediatric center in South Vietnam. The patient was considered feasible if he (or she) did not have the contra-indication for the ketogenic diet
  Interventions: Dietary Supplement: Ketogenic diet
- the tolerability of the ketogenic diet (Experimental): The purpose of this study was to verify the tolerability of the ketogenic diet in children with refractory epilepsies followed at a pediatric center in South Vietnam. The patient was considered tolerant if he (or she) did not have any side effects caused by the ketogenic diet
  Interventions: Dietary Supplement: Ketogenic diet
- the efficacy of the ketogenic diet (Experimental): The purpose of this study was to verify the efficacy of the ketogenic diet in children with refractory epilepsies followed at a pediatric center in South Vietnam. Patients were considered responders when a 50% seizure frequency was reached.
  Interventions: Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — The ketogenic diet (KD) has been shown as an effective alternative for patients with drug-resistant epilepsy

SUMMARY:
According to the World Health Organization, more than 50 million people have epilepsy. Among them, nearly 80% of epileptic patients live in developing countries and 75% of them do not have access to treatment. The ketogenic diet (KD) has been shown as an effective alternative for patients with drug-resistant epilepsy. Although it has been studied by few studies in Asia, no such studies have been conducted in Vietnam. The purpose of this study was to verify the feasibility, tolerability, and efficacy of the KD in children with refractory epilepsies followed at a pediatric center in South Vietnam.

DETAILED DESCRIPTION:
Children with drug-resistant epilepsy followed at Children's Hospital No.2, Viet Nam treated by KD were included in a prospective study from June 2019 to October 2021. Side-effects, retention rate, number, and duration of seizures were recorded after 1, 3, 6, 9, and 12 months of KD. Patients were considered as responders when a 50% seizure frequency was reached. Tolerance and acceptability of the KD were closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* age from 1 to 10 years at the time of enrolment,
* drug-resistant epilepsy according to the 2010 ILAE criteria,
* an indication for a ketogenic diet trial according to the 2018 ILAE recommendations

Exclusion Criteria:

- clinical or laboratory features suggesting an underlying disease contra-indication the use of a ketogenic diet

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
The feasibility of the ketogenic diet | 12 months
  Number of drug-resistant epilepsy patients without ketogenic diet's contra-indication
The tolerability of the ketogenic diet at 12 months | 12 months
  Number of participants without ketogenic diet's side effect at 12 months
The efficacy of the ketogenic diet at 12 months | 12 months
  The number of participants had a 50% seizure decrease at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- N02 Children's Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No